CLINICAL TRIAL: NCT02570347
Title: Routine vs. Clinically-Directed Antibiotic Treatment in Snake Bite With Local Envenomation: a Randomised Controlled Trial
Brief Title: Routine Antibiotic vs. Directed Antibiotic Treatment in Snake Bite
Acronym: RADIANS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slower than anticipated recruitment and emergent COVID-19 situation
Sponsor: Jawaharlal Institute of Postgraduate Medical Education & Research (Other Government)
Responsible Party: Principal Investigator, Tamilarasu Kadhiravan, MD, Professor of Medicine, Jawaharlal Institute of Postgraduate Medical Education & Research
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JIP/IEC/2015/17/649
Record Dates: First submitted 2015-10-05; First posted 2015-10-07 (Estimated); Last update posted 2025-05-30 (Actual); Status verified 2025-05

CONDITIONS: Snake Bites
Keywords: Snake Envenomation; Antibiotic Prophylaxis; Viperidae
MeSH Terms: conditions — Snake Bites | interventions — Amoxicillin-Potassium Clavulanate Combination; Tetanus Toxoid

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Routine use arm (Active Comparator): All participants allocated to this arm will be given
  * Injection Tetanus toxoid 0.5 ml intramuscularly Stat
  * Antibiotic (Co-amoxiclav) will be given to all patients for a minimum duration of 5 days.
  * Daily clinical assessment would be done. Change of antibiotics is allowed if clinical failure occurs.
  Use of antibiotics for emergent indications unrelated to the bitten limb such as nosocomial infections would be allowed at the treating physician's discretion.
  Interventions: Drug: Co-amoxiclav; Biological: Tetanus toxoid
- Clinically-directed use arm (Experimental): Participants allocated to this arm will be given
  * Injection Tetanus toxoid 0.5 ml intramuscularly Stat
  * Daily clinical assessment would be done. Antibiotic (Co-amoxiclav) will be started only if clinical failure occurs.
  Use of antibiotics for emergent indications unrelated to the bitten limb such as nosocomial infections would be allowed at the treating physician's discretion.
  Interventions: Drug: Co-amoxiclav; Biological: Tetanus toxoid

INTERVENTIONS:
Drug: Co-amoxiclav — Injection Co-amoxiclav 1.2 g intravenously q8h for a minimum of 48-72 hours; switched to oral Co-amoxiclav 625 mg b.i.d. when clinically appropriate.
  Other Names: Augmentin
Biological: Tetanus toxoid — Injection Tetanus toxoid 0.5 ml intramuscularly Stat

SUMMARY:
Clinicians tend to overuse antibiotics in snake bite despite evidence from three previous clinical trials that failed to show a benefit. But, none of these trials was done in India. Further, the species of snake in two of these trials was quite different from that seen in the Indian setting limiting generalization of these findings. Hence, home-grown evidence is needed to persuade clinicians to use antibiotics rationally.

DETAILED DESCRIPTION:
Snake bite is a common clinical problem in India and elsewhere, affecting agricultural workers and rural population, resulting in thousands of deaths every year. Apart from causing systemic manifestations such as coagulopathy, acute renal failure, and neuroparalysis, local effects of the venom manifest as swelling of the bitten limb. Despite administration of adequate antivenom, the limb swelling progresses in the first 48-72 hours accompanied by considerable pain. Often the limb swelling is accompanied by formation of blebs and gangrenous skin changes. At times, the limb swelling is severe enough to result in compartment syndrome, necessitating surgical interventions such as fasciotomy and debridement. Animal bites are typically associated with a risk of infection by the oral flora. Likewise, apart from releasing the venom, inoculation of oral flora as a result of snake bite could result in local infectious complications adding to the deleterious effects of the snake venom.

Observational studies suggest that the risk of infection following simple bites on the lower limbs is much less than what is often believed, and evidence from clinical trials also does not support routine use of antibiotics in snake bite. For this reason, clinical practice guidelines do not recommend routine prophylactic use of antibiotics in snake bite. But, in reality, many clinicians continue to use antibiotics routinely in all venomous snake bites hoping to prevent a local infection. While such a strategy may not reduce the risk of infection, it would result in overuse of antibiotics promoting antimicrobial resistance and escalating treatment costs.

The investigators hypothesize that clinically-directed use of antibiotics would be non-inferior to routine use in preventing local infectious complications of snake bite, while being superior in reducing the antibiotic consumption. Non-inferiority would be inferred if the one-sided 95% CI of the difference does not exceed 10% in favour of the routine use arm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years
* History of snake bite with features of local envenomation with/without systemic features
* Less than 24 hours since bite, AND
* No prior antibiotic treatment

Exclusion Criteria:

* Upper limb bites
* Multiple (> 1) bites
* Wound manipulation
* Extensive local necrosis or blebs
* Seriously-ill patients with hypotension/capillary leak/life threatening bleeding.
* Suspected cobra bite, OR
* Pregnant/breast-feeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2016-05-03 (Actual); Primary Completion 2019-10-24 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Clinical failure | up to 4 weeks
  Defined as occurrence of any one of the following on daily assessments - Abscess formation at any point of time; Surgical debridement/fasciotomy at any time; Worsening limb swelling beyond 72-96 hours or appearance of necrosis or blebs along with any one of the following: fever, persistent or worsening leucocytosis, or global deterioration on clinical assessment.
Antibiotic consumption | up to 4 weeks
  Defined as the total amount of all antibiotics consumed regardless of clinical indication expressed in terms of defined daily doses (DDD).

SECONDARY OUTCOMES:
Length of hospital stay | up to 4 weeks
  Number of days from hospital admission until discharge
Anti-snake venom consumption | up to 4 weeks
  The total number of vials of the anti-venom administered including doses received prior to being brought to JIPMER.
New-onset organ failure | up to 4 weeks
  This includes acute kidney injury (AKI) defined as peak serum creatinine > 2 mg/dL, shock defined as systolic blood pressure < 90 mm Hg requiring use of vasopressors; bleeding from any site necessitating transfusion of blood/blood products; and capillary leak syndrome.
Death/need for surgical intervention | up to 4 weeks
  This would be a composite measure of death and/or need for surgical intervention. Death indicates in-hospital death due to any cause during the index hospitalisation. Surgical intervention would include need for any surgical intervention such as incision and drainage of abscess, wound debridement for necrosis or gangrene, fasciotomy for compartment syndrome, etc.
Drug-related adverse events | up to 4 weeks
  Any suspected or confirmed adverse drug reaction

CONTACTS AND LOCATIONS:
Overall Officials: Tamilarasu Kadhiravan, M.D., Principal Investigator — Jawaharlal Institute of Postgraduate Medical Education & Research
Locations (1):
- Department of Medicine, Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry, Puducherry, India

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data that underlie the published results (text, tables, figures and appendices).
Supporting Information: Study Protocol, ICF, CSR
Time Frame: Immediately following publication for up to 5 years.
Access Criteria: Anyone who wishes to access the data, upon reasonable request to the principal investigator.
URL: https://bmjopen.bmj.com/

REFERENCES:
- [Background] Terry P, Mackway-Jones K. Towards evidence based emergency medicine: best BETs from the Manchester Royal Infirmary. The use of antibiotics in venomous snake bite. Emerg Med J. 2002 Jan;19(1):48-9. doi: 10.1136/emj.19.1.48. PMID 11777875
- [Background] Terry P, Mackway-Jones K. Towards evidence based emergency medicine: best BETs from the Manchester Royal Infirmary. Antibiotics in non-venomous snakebite. Emerg Med J. 2002 Mar;19(2):142. doi: 10.1136/emj.19.2.142. PMID 11904264
- [Background] Jorge MT, Malaque C, Ribeiro LA, Fan HW, Cardoso JL, Nishioka SA, Sano-Martins IS, Franca FO, Kamiguti AS, Theakston RD, Warrell DA. Failure of chloramphenicol prophylaxis to reduce the frequency of abscess formation as a complication of envenoming by Bothrops snakes in Brazil: a double-blind randomized controlled trial. Trans R Soc Trop Med Hyg. 2004 Sep;98(9):529-34. doi: 10.1016/j.trstmh.2003.12.009. PMID 15251401
- [Background] Kularatne SA, Kumarasiri PV, Pushpakumara SK, Dissanayaka WP, Ariyasena H, Gawarammana IB, Senanayake N. Routine antibiotic therapy in the management of the local inflammatory swelling in venomous snakebites: results of a placebo-controlled study. Ceylon Med J. 2005 Dec;50(4):151-5. doi: 10.4038/cmj.v50i4.1405. PMID 16538909
- [Background] Kerrigan KR, Mertz BL, Nelson SJ, Dye JD. Antibiotic prophylaxis for pit viper envenomation: prospective, controlled trial. World J Surg. 1997 May;21(4):369-72; discussion 372-3. doi: 10.1007/pl00012255. PMID 9143566
- [Background] Mohapatra B, Warrell DA, Suraweera W, Bhatia P, Dhingra N, Jotkar RM, Rodriguez PS, Mishra K, Whitaker R, Jha P; Million Death Study Collaborators. Snakebite mortality in India: a nationally representative mortality survey. PLoS Negl Trop Dis. 2011 Apr 12;5(4):e1018. doi: 10.1371/journal.pntd.0001018. PMID 21532748
- [Derived] Gautam A, Indu MB, Bhardwaj A, Sabitha P, Deepanjali S, Suryanarayana BS, Bammigatti C, Kadhiravan T. Clinically directed initiation versus routine use of amoxicillin-clavulanate and the risk of local complications among patients with haemotoxic snakebite envenomation treated at a teaching hospital in southern India: a randomised, non-inferiority trial. BMJ Open. 2025 Jun 23;15(6):e094409. doi: 10.1136/bmjopen-2024-094409. PMID 40550712